CLINICAL TRIAL: NCT02759549
Title: Fatigue in Breast Cancer Patients Undergoing Radiotherapy-Electronic Self-Management Resource Training for Mental Health (eSMART-MH)
Brief Title: Fatigue in Breast Cancer Patients Undergoing Radiotherapy-eSMART-MH
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Principal Investigator, Mylin Torres, MD, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00028295
Record Dates: First submitted 2016-04-29; First posted 2016-05-03 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Breast Cancer
Keywords: Radiation Therapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- eSMART-MH (Experimental): Participants undergoing radiation treatment for breast cancer will receive the Electronic Self-Management Resource Training for Mental Health (eSMART-MH) intervention.
  Interventions: Behavioral: eSMART-MH; Other: Mobile Mood Tracking (Mood 24/7)
- Theater Testing (Other): Participants undergoing radiation treatment for breast cancer will participate in a theater testing workshop.
  Interventions: Behavioral: Theater Testing Workshop

INTERVENTIONS:
Behavioral: eSMART-MH — eSMART-MH (Electronic Self-Management Resource Training for Mental Health) is a software, which is set in a 3-D virtual primary care office environment in which a subject interacts with avatar virtual healthcare staff (medical receptionist, medical assistant, providers, and a virtual healthcare coach). The avatars are programmed to behave like humans. The subject moves through the 3-D virtual primary care office and encounters virtual healthcare staff and providers. The subject practices discussing depressive symptoms with avatar healthcare providers and practices self-management skills related to symptoms of depression.The subject also interacts with the health care coach. The health care coach provides the subject with real-time strategies to enhance communication with healthcare providers during their virtual office visit. eSMART-MH will be used once a week throughout the duration of radiation treatment.
  Arms: eSMART-MH
Other: Mobile Mood Tracking (Mood 24/7) — Public social media data posted by participants will be accessed and downloaded to a computer program. Permission for the study team to access this data is optional.
  Arms: eSMART-MH
Behavioral: Theater Testing Workshop — The theater testing workshop consists of one to two one-on-one sessions with study staff during which participants will review a computer program for its content and usability, as well as discuss areas for improvement. Participants will also be asked to complete questionnaires and a attend a brief interview regarding any suggested improvements for the computer program.
  Arms: Theater Testing

SUMMARY:
The purpose of this study is to determine if an avatar-based depression self-management intervention (eSMART-MH) once a week for the duration of the participant's radiation treatment will significantly reduce depressive symptoms. Investigators also seek to explore how women with breast cancer describe their mood using prompted and unprompted speech through electronic social media and interviews.

Participants will be randomized into the eSMART-MH group or the theater testing (attention control) group. In addition to the assigned interventions, participants will be asked to complete questionnaires and interviews with the study staff.

DETAILED DESCRIPTION:
The purpose of this study is to determine if an avatar-based depression self-management intervention (eSMART-MH) once a week for the duration of the participant's radiation treatment will significantly reduce depressive symptoms. Investigators also seek to explore how women with breast cancer describe their mood using prompted and unprompted speech through electronic social media and interviews.

Participants will be randomized into the eSMART-MH group or the theater testing (attention control) group. In addition to the assigned interventions, participants will be asked to complete questionnaires and interviews with the study staff.

Participants will be enrolled within two weeks of radiotherapy. A preliminary depression survey (IDS-SR) will be given to assess depression. There will be a total of three routine study assessments, one within two weeks prior to the beginning of radiotherapy, one the last week of radiotherapy and one 5 - 7 weeks after radiotherapy is completed.

ELIGIBILITY:
Inclusion Criteria:

* Patients seen in the Emory Breast Center at The Emory Clinic and Emory Midtown Hospital who are treated with curative intent.
* Score of 8 or higher on the Inventory of Depressive Symptomology - Self Reported (IDS-SR) test

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change in an Inventory of Depressive Symptomatology-Self Reported (IDS-SR) score | Baseline, Post Treatment (5-7 weeks)
  The IDS-SR is a self-reported measure in which participants rate the frequency of depression symptoms within the past seven days. Scores range from 0 to 84, with higher score reflecting greater severity of depressive symptoms.

SECONDARY OUTCOMES:
Change in Pittsburgh Sleep Quality Index (PSQI) Score | Baseline, Post Treatment (5-7 weeks)
  The PSQI is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. Scores range from 0 to 21. A score of less than or equal to 5 is associated with good sleep quality. A score greater than 5 is associated with poor sleep quality.
Change in Perceived Stress Scale (PSS) Score | Baseline, Post Treatment (5-7 weeks)
  The PSS is a self-reported instrument used to measure the perception of stress. Scores range from 0 to 40. Score of 20 or higher are considered high stress.
Change in Short Form-36 (SF-36) Health Survey Score | Baseline, Post Treatment (5-7 weeks)
  The SF-36 is a self-reported survey of health status. Scores range from 0 to 100. Lower scores indicate disability. The higher the score, the less disability.
Change in Godin Leisure-Time Exercise Questionnaire (GLTEQ) Score | Baseline, Post Treatment (5-7 weeks)
  The GLTEQ is a self-reported questionnaire used to measure usual leisure-time exercise habits during a typical seven day period. A score of 24 or more indicates active and substantial exercise benefits. A score of 23 units or less indicates insufficiently active and less substantial exercise benefits.
Change in Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue Short Form Score | Baseline, Post Treatment (5-7 weeks)
  The PROMIS Fatigue questionnaire is a self-report tool used to evaluate frequency, duration, and intensity of fatigue over the past seven days. Scores range from 7 to 35. The higher the score, the more fatigue.
Change in Lent Soma Scale Patient Questionnaire Score | Baseline, Post Treatment (5-7 weeks)
  The Lent Soma questionnaire is a self-reported measure of pain. Scores range from 0 to 9. The higher the score, the more pain reported.
Change in Multidimensional Fatigue Inventory (MFI) Score | Baseline, Post Treatment (5-7 weeks)
  The Multidimensional Fatigue Inventory (MFI) is a 20-item self-report instrument designed to measure fatigue. Scores range from 20 to 100.The higher the score, the more fatigued.
Change in The Centers for Disease Control (CDC) Health-Related Quality of Life-4 (QOL) Questionnaire Score | Baseline, Post Treatment (5-7 weeks)
  Quality of Life will be measured by the Center for Disease Control Health Related Quality of Life-4 (CDC HRQOL). This self-report measures quality of life over the last 30 days in the domains of physical and mental health.
Change in Functional Assessment of Cancer Therapy-General (FACT-G) Score | Baseline, Post Treatment (5-7 weeks)
  The FACT-G is a self-reported measure of well being in the past seven days. Scores range from 0 to 27. A higher score indicates worse perception of well being.

OTHER OUTCOMES:
Change in Behavioral Activation for Depression Scale-Short Form (BADS-SF) Score | Baseline, Post Treatment (5-7 weeks)
  The BADS-SF is a 9-item self-report measures that assess behavioral activation which captures the domains of activation, avoidance/rumination, work/school impairment, and social impairment. The BADS-SF asks participants to respond to each statement over the past week, including the day in which they complete the measure, on a 0 to 6 likert type scale.The BADS-SF has shown to be significantly associated with depression.
Change in Self-Efficacy for Managing Chronic Disease 6-Item Scale Score | Baseline, Post Treatment (5-7 weeks)
  The Self-Efficacy for Managing Chronic Disease questionnaire is a six item self-report scale. This measure asks how confident, on a scale of 1-10, the respondent is in doing certain activities pertaining to self-management. Scores range from 6 to 60. A higher score indicates more confidence.
Change in Pediatric CARE measure 10 questions (PCM 10Q) Score | Baseline, Post Treatment (5-7 weeks)
  The PCM 10Q is used to gain the views of children or patients receiving health services. It is a patient-centered measure of relational empathy. It measures patients' experiences of the interpersonal aspects of clinical encounters.
Change in Virtual Support Measure Score | Baseline, Post Treatment (5-7 weeks)
  The virtual support questionnaire is a measure of perceived virtual support of the avatars. Participants rate the "virtual support" provided by the avatar healthcare provider and avatar coach separately. The first 12 questions of the Virtual Support Questionnaire ask participants to rate, on a Likert-type format, the avatars on a variety of relational characteristics. Selection options range from (1) "No, not at all" to (5) "Yes, definitely." The last 10 items of the Virtual Support Questionnaire ask respondents to rate, using a Likert-type format, to what degree they agree or disagree with statements about how the avatars understood their experiences. Selection options ranged from (1) "Strongly agree" to (6) "Strongly disagree."
Change in The University of California, Los Angeles (UCLA) Loneliness Scale Score | Baseline, Post Treatment (5-7 weeks)
  The UCLA Loneliness Scale is a 20-item scale designed to measure one's subjective feelings of loneliness as well as feelings of social isolation. Participants rate each item as either O ("I often feel this way"),S ("I sometimes feel this way"), R ("I rarely feel this way"), N ("I never feel this way"). A higher score indicates more feelings of loneliness.This scale has a strong association with depression.
Change in Patient Activation Measure (PAM-13) Score | Baseline, Post Treatment (5-7 weeks)
  The PAM-13 is a 13-item measure that assesses the patient's perception of their knowledge, skill, and confidence in self-management behavior. Scores range from 0-100, with a higher score indicating greater patient activation.
Change in Quality of Patient-Provider Interaction Questionnaire (QPPI) Score | Baseline, Post Treatment (5-7 weeks)
  The QPPI is a 14-item self-report likert type style questionnaire that assesses from the patient's perspective the quality of the interaction between the patient provider.
Change in Patient Self-Competence Subscale (PSCS) Score | Baseline, Post Treatment (5-7 weeks)
  A 16-item five point Likert scale that asks participants to rate items from 5 (important) to 1 (unimportant); a higher score indicates greater perceived self-competence and effective communication with a health care provider.
Change in FAS Verbal Fluency Test Score | Baseline, Post Treatment (5-7 weeks)
  The FAS Verbal Fluency Test task asks respondents to generate words beginning with the letters "F," "A," and "S" within 60 seconds. Adults with depression generate fewer words on the FAS than non-depressed.
Change in The State Hope Scale Score | Baseline, Post Treatment (5-7 weeks)
  The State Hope Scale is a a 6-item self-report scale which measures goal-directed thinking and the "here and now." Respondents are asked to respond to items in relation to what is "going on in your life right now" in response to goal-directed statements on a 1-8 scale.
Change in Emotional Regulation Questionnaire (ERQ) Score | Baseline, Post Treatment (5-7 weeks)
  The ERQ is a 20-item scale that asks respondents how they manage and regulate their emotions in response to life events on a 1-7 likert-type scale.
Change in Body Awareness Questionnaire Score | Baseline, Post Treatment (5-7 weeks)
  The Body Awareness Questionnaire is a an 18-item measure that asks respondents to rate their sensitivity to normal and non-emotional body processes on a 1-7 likert-type scale.
Change in Experiences Questionnaire (EQ) Score | Baseline, Post Treatment (5-7 weeks)
  The EQ is a 20 item self-report scale designed to measure decentering and deep thinking.
3 Item Functional Health Literacy Quick Screen | Baseline
  The 3 Item Functional Health Literacy Quick Screen is used to detect limited and marginal health literacy skills.
Tobacco Use Questionnaire | Baseline
  The Tobacco Use Questionnaire is two question self-report about the use of traditional cigarettes, or e-cigarettes, or both and the amount of cigarettes smoked.
Alcohol Use Disorders Identification Test (AUDIT) | Baseline
  The AUDIT simple brief assessment tool to screen for excessive drinking. The measure consists of 10 questions about recent alcohol use, alcohol dependence symptoms, and alcohol-related problems.
Adverse Childhood Event (ACE) Questionnaire | Post last intervention (4 week follow up)
  An ACE score is a tally of different types of abuse, neglect, and household dysfunction. There are 10 items on the measure; we will ask 9 of these questions, omitting the question about sexual abuse. The ACE Study emphasizes the number rather than categories of ACE that one has been subjected to. The number of the nine items of ACE that one has undergone (0-9) is regarded as the ACE score.

CONTACTS AND LOCATIONS:
Overall Officials: Mylin Torres, MD, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - Emory Clinic, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Winship Cancer Institute, Atlanta, Georgia